CLINICAL TRIAL: NCT04806932
Title: Comparison of the Modified Approach and Conventional Approach of Radial Artery Cannulation Under Short-axis Ultrasound Guidance in Intensive Care Unit(ICU) Hypotensive Patients: a Randomized Controlled Study.
Brief Title: Comparison of the Modified and Conventional Approach of Radial Artery Cannulation Under Short-axis Ultrasound Guidance in ICU Hypotensive Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Yangpu District Central Hospital Affiliated to Tongji University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MARS
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-03

CONDITIONS: Radial Artery Catheterization
Keywords: radial artery catheterization, ultrasound, hypotensive, critical ill

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients were randomized to the conventional Approach (CA) or modified Approach (MA) group in a 1:1 ratio using a computerized system. The allocation process was intensively managed by an allocation group using sequentially numbered containers and the allocation result was concealed until it was implemented. When a patient was eligible, the investigator informed the allocation group to get intervention group allocated to the patient: CA orMA group. Because of feasibility issues, operators were not blinded to the assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The modified approach (Active Comparator): The first three attempts via the modified approach will be performed. If the first three attempts failed, the location or operator of the subsequent attempts of artery puncture will be changed.
  Interventions: Procedure: The modified approach
- The conventional approach (Placebo Comparator): The first three attempts via the conventional approach will be performed. If the first three attempts failed, the location or operator of the subsequent attempts of artery puncture will be changed.
  Interventions: Procedure: The conventional approach

INTERVENTIONS:
Procedure: The modified approach — The first three attempts via the modified approach will be performed. If the first three attempts failed, the location or operator of the subsequent attempts of artery puncture will be changed.
  Arms: The modified approach
Procedure: The conventional approach — The conventional approach
  Arms: The conventional approach

SUMMARY:
Radial artery cannulation can be performed under short-axis ultrasound guidance. However, the first puncture success rate was low in patients with hypotensive patients. Compared with the conventional approach, the modified approach combined the ultrasonic location system with a dynamic needle tip positioning technique. The aim of our study is to compare the first puncture success rate and safety between the two approaches of ultrasound-guided radial artery cannulation in hypotensive ICU patients.

DETAILED DESCRIPTION:
Hypotensive patients in the intensive care unit may have extremely unstable hemodynamics. Blood pressure is the most important outcome in the diagnosis and treatment of shock. Vasopressor drugs are often required to maintain blood pressure in addition to fluid infusion. Noninvasive blood pressure measurement is unable to meet the clinical requirements. It is necessary to establish an invasive blood pressure monitoring method as soon as possible that can observe the real-time pressure. Radial artery cannulation has become the most commonly used due to its superficial location and less severe complication. However, radial artery cannulation is difficult to achieve in hypotensive patients due to weak radial artery pulsation, small arterial diameter, and peripheral vasospasm as blood flow is directed toward central vessels.

Some studies have shown that ultrasound-guided cannulation is more successful than the palpation technique. However, the success rate is largely dependent on the ultrasound operator's experience and skills. The operator requires good hand-eye coordination, technical skills, and some experience to overcome this shortcoming of ultrasound, which limits the advantages of ultrasound-guided vascular puncture, especially for operators with insufficient experience. There are 2 basic approaches in needling techniques: short-axis out-of-plane(SA-OOP) and long-axis in-plane(LA-IP) techniques.

In-plane technology requires the operator to be very skilled at ultrasound technology, which is more dependent on experience and can be difficult for novices to master; on the other hand, given that the long axis is subject to slice-thickness artifacts, due to the measurable thickness of the ultrasound beam itself, the cannula in the long axis appears to be in the same plane as the extremely small radial artery, even when the cannula has not been successfully inserted into the artery. Therefore, we prefer the out-of-plane technique.

The short-axis view has the advantages of providing better visualization of the surrounding structures and easier imaging which is convenient for novices to master. The procedure of radial artery puncture can be divided into 3 steps. The first step is to locate the puncture site, the second step is the puncture, and the last step entails the insertion of the cannula into the radial artery.

The first step is particularly important because appropriate localization facilitates the success of the puncture and insertion. The first difficulty encountered during radial artery puncture is the exact positioning of the puncture point. Ultrasound with developing lines guided by dynamic ultrasound has achieved a good effect in patients without hypotension. In the group with the modified technique, we use the developing line to locate the puncture site.

The second difficulty encountered during radial artery puncture is the risk of posterior wall penetration. With the dynamic needle tip positioning(DNTP) technique, the operator keeps real-time track of the position of the needle tip at all times which significantly reduces the chance of posterior wall perforation. We combined the developing line and DNTP technique in the modified group and assume that the technique theoretically increases the success rate and decreases the complication rate of radial artery puncture. Therefore, in this trial, we compared the success rate of radial artery puncture using the traditional method and modified technique in hypotensive ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients in intensive care units;
* The need for invasive hemodynamic monitoring (arterial blood pressure and cardiac output monitoring);
* The need for frequent blood sampling (arterial blood gas analysis and general laboratory evaluation);
* Vasopressor therapy;

Exclusion Criteria:

* a negative Allen test;
* ulnar artery occlusion;
* prevalent atherosclerosis;
* a blocked or embolized target vessel determined by ultrasound assessment;
* Raynaud disease;
* infection near the radial artery puncture site;

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2021-04-11 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
First-pass success | approximately 3 minutes
  successful catheterization on the first attempt

SECONDARY OUTCOMES:
Overall success | within 10 minutes
  successful catheterization without a limit on the number of punctures.
The cannulation time | within 10 minutes
  the interval between skin contact with the probe and confirmation of the arterial waveform on the monitor.
Posterior wall puncture | within 10 minutes
  the operator saw the needle passing the posterior wall or blood backflow appeared then disappeared while needle advancing.
the number of attempts | within 10 minutes
  the number of attempts until successful cannulation
Complication rate | Day 1
  bleeding, hematoma,thrombosis, vasospasm, occlusion, aneurysm

CONTACTS AND LOCATIONS:
Overall Officials: Guowei Tu, PhD, Principal Investigator — Fudan University
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quan Z, Tian M, Chi P, Cao Y, Li X, Peng K. Modified short-axis out-of-plane ultrasound versus conventional long-axis in-plane ultrasound to guide radial artery cannulation: a randomized controlled trial. Anesth Analg. 2014 Jul;119(1):163-169. doi: 10.1213/ANE.0000000000000242. PMID 24806143
- [Background] Liu L, Tan Y, Li S, Tian J. "Modified Dynamic Needle Tip Positioning" Short-Axis, Out-of-Plane, Ultrasound-Guided Radial Artery Cannulation in Neonates: A Randomized Controlled Trial. Anesth Analg. 2019 Jul;129(1):178-183. doi: 10.1213/ANE.0000000000003445. PMID 29787409
- [Background] Clemmesen L, Knudsen L, Sloth E, Bendtsen T. Dynamic needle tip positioning - ultrasound guidance for peripheral vascular access. A randomized, controlled and blinded study in phantoms performed by ultrasound novices. Ultraschall Med. 2012 Dec;33(7):E321-E325. doi: 10.1055/s-0032-1312824. Epub 2012 Oct 11. PMID 23059741